CLINICAL TRIAL: NCT05395156
Title: EFFECT OF TENS ON ACUPOINTS IN PREMENSTRUAL SYNDROME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aml Mohammed Elsayed Abdelaal, spicialist of physical therapy at talkha central hospital, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003688
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Premenstrual Pain
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham acupoint (Experimental): Control group: (placebo group) will be consisted of twenty-five females diagnosed with premenstrual syndrome. They will receive TEAS on sham acupoint (the acupoint selection site was 1 inch away from the acupoint selection in the study group) daily from 3 days before menstruation to the 4th day of menstruation for 3 consequent menstrual cycles with average of 7 sessions per month for 3 months
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Electroacupuncture (Experimental): Study group: (Electroacupuncture group) will be consisted of twenty-five females diagnosed with premenstrual syndrome. They will receive TEAS on neurogenic acupoints daily from 3 days before menstruation to the 4th day of menstruation for 3 consequent menstrual cycles with average of 7 sessions per month for 3 months.
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Control group will receive TEAS on sham acupoint daily from 3 days before menstruation to the 4th day of menstruation for 3 consequent menstrual cycles Study group will receive TEAS on neurogenic acupoints daily from 3 days before menstruation to the 4th day of menstruation for 3 consequent menstrual cycles

SUMMARY:
These will be no effect of transcutaneous electrical acupoint stimulation on premenstrual syndrome Does transcutaneous electrical acupoint stimulation affect premenstrual syndrome (PMS)?

DETAILED DESCRIPTION:
Premenstrual syndrome is a collection of emotional, physiological, and behavioral symptoms that develop around the end of the luteal phase and fade away with or after menstruation Due to limited evidence on the efficacy of sustained progesterone and the side effects of antidepressant and anxiolytics, in some cases, alternative therapies are recommended for patients with PMS TEAS may be more effective than other forms of transcutaneous electrical nerve stimulation (TENS) in modulating brain activity because acupoint areas contain relatively denser neural and neuroactive components than non-acupoint areas TEAS has been reported to have similar efficacy as acupuncture, electrical acupuncture, and TENS

ELIGIBILITY:
Inclusion Criteria:

* Their age will range from 18 to 25 years.
* The regularity of menstrual cycle is 28-35 days.
* All of them suffering from moderate and sever PMS.
* All participants are virgin.
* Their BMI will range from 25-30 kg\m2.

Exclusion Criteria:

* Any pathological findings in the pelvic cavity as PCO, Endometriosis and pelvic inflammatory disease.
* Any history of gynecological intervention.
* Have any condition impedes the use of electrotherapy.
* Receiving sedatives or any medical treatment.
* Having irregular menstruation.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-10 (Estimated); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
pain severity | Up to 3 monthes
  The pain intensity will be assessed through visual analogue scale (VAS) for each participant in both groups before and after treatment Each participant will be asked to mark a point on VAS line between the extremes that related to her current pain intensity
premenstrual syndrome severity | up to 3 monthes
  Participants can differentiate between their experiences of different symptoms during menstrual cycle and they will be assessed before and after treatment using the Menstrual Distress Questionnaire (MDQ) Each participant will be asked to rate their experience of each of the symptoms on the MDQ on a scale ranging from no experience of the symptom to an acute or partially disabling experience of the symptom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF